CLINICAL TRIAL: NCT05231408
Title: Effects of High-Intensity Interval Aerobic Exercise Training on Oxygen Consumption Muscle Oxygenation and Physical Activity Level in Patients With Post COVID-19
Brief Title: Effects of Aerobic Exercise in Patients With Post COVID-19
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Study director, PT, PhD, Prof.Dr. Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Head of Cardiopulmonary Rehabilitation Clinic, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Gazi University 90
Record Dates: First submitted 2022-02-08; First posted 2022-02-09 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: COVID-19
Keywords: COVID-19; aerobic exercise training; muscle oxygenation; oxygen consumption; physical activity
MeSH Terms: conditions — COVID-19; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple-blind study; the patients will not be informed about their groups (training group or the control group) and they will be evaluated and trained at different places and times.
  Evaluations and interventions will be performed different physiotherapist. In addition, before statistical analysis patients' groups will be coded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental): Training group will receive high-intensity interval aerobic exercise training on treadmill accompanied by physiotherapist for 8 weeks.
  Interventions: Other: High-intensity interval aerobic exercise training
- Control Group (Sham Comparator): Breathing exercises will be given to control group as a home program for 8 weeks.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: High-intensity interval aerobic exercise training — High-intensity interval aerobic exercise training will be given to training group on treadmill 3 days in a week and 15-45 minutes in a day for 8 weeks with the assistance of a physiotherapist.
  The training workload of the active phase of high-intensity interval aerobic exercise training will be applied at 80-100% of peak oxygen consumption or 85-95% of peak heart rate or according to Borg scale dyspnea/fatigue 15-18 points.
  The training workload of the active recovery phase of high-intensity interval aerobic exercise training will be applied at 50-60% of peak oxygen consumption or 60-75% of peak heart rate or according to Borg scale dyspnea/fatigue 11-13 points.
  Arms: Training Group
Other: Control Group — Breathing exercises will be given to the control group 120 times in a day and 7 days in a week for 8 weeks as a home program. The control group will be followed-up by telephone once a week.
  Arms: Control Group

SUMMARY:
Many structures and organs are adversely affected after COVID-19. The most obvious and common problem is lung involvement. In the pathology report of the patients, it has been shown that there are changes such as diffuse alveolar damage, bronchiolitis and interstitial fibrosis. The most prominent effect of COVID-19 in patients with reduced lung functions is reduced diffusion capacity. While the disease severity worsens, pulmonary fibrosis becomes more pronounced in cases. The complaints of dyspnea and fatigue of patients after discharged continue. Inspiratory and expiratory respiratory muscle weakness are observed in more than 50% of patients with COVID-19, measured in the first month after the discharged. This respiratory muscle weakness is associated with myopathy due to hypoxemia, oxygen support, prolonged bed rest and corticosteroid use, regardless of disease severity.

It is seen that these patients with COVID-19 need exercise training because of lung involvement, decreased exercise capacity and persistence of some symptom complaints after the discharged.

DETAILED DESCRIPTION:
Patients with COVID-19 have not only reduced respiratory capacity, but also diminished muscle strength, exercise capacity, weakness cardiac system. In parallel with aforementioned, physical activity level and quality of life get worse in this patients. Therefore, the patients with COVID-19 need exercise training after the discharged. In the literature, the achievement of exercise training in many aspects such as exercise capacity, lung health, respiratory muscle strength, dyspnea has been proven in many diseases such as chronic obstructive pulmonary disease and heart failure.

Effects of high-intensity interval aerobic exercise training on oxygen consumption, muscle oxygenation, physical activity level, pulmonary function, functional exercise capacity, respiratory and peripheral strength, inspiratory muscle endurance, functional status, dyspnea, fatigue perception and quality of life have not been investigated in literature in patients with COVID-19. According to inclusion and exclusion criteria, 15 patients for training group and 15 patients for control group will be included. All assessments will be completed in two days before and after eight weeks training.

Primary outcome measurement will be oxygen consumption (cardiopulmonary exercise test).

Secondary outcome will be muscle oxygenation (Moxy device), physical activity level (multi sensor activity device), pulmonary function (spirometer), functional exercise capacity (six-minute walk test), respiratory (mouth pressure device) and peripheral muscle (hand-held dynamometer) strength, inspiratory muscle endurance (incremental threshold loading test), functional status (Post-COVID-19 Functional Status Scale), dyspnea (London Chest Daily Living Activity Scale), fatigue (Fatigue Severity Scale) and quality of life (Saint George Respiratory Questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* aged between 18-75 years
* diagnosed with COVID-19 before
* patients whose COVID-19 Polymerase Chain Reaction test turned negative or be negative already
* patients who are willing to participate in this study

Exclusion Criteria:

Patients with

* body mass index >35 kg/m2
* cancer, renal or hepatic diseases
* aortic stenosis, complex arrhythmia, aortic aneurysm
* serious neurological, neuromuscular, orthopedic, other systemic diseases or other diseases affecting physical functions
* uncontrolled hypertension and/or diabetes mellitus, heart failure and cardiovascular disease
* acute pulmonary exacerbation, acute upper or lower respiratory tract infection
* cognitive impairment that causes difficulty in understanding and following exercise test instructions
* bulla formation in the lung
* participated in a planned exercise program in the last three months
* contraindication for exercise testing and/or exercise training according to the American College of Sports Medicine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-25 (Actual); Primary Completion 2024-08-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Oxygen consumption | First day
  Maximal exercise capacity will be assessed with symptom limited cardiopulmonary exercise test on a treadmill at a progressively increasing speed and grade. Oxygen consumption will be measured during the test.

SECONDARY OUTCOMES:
Muscle Oxygenation | First and second day
  Muscle oxygenation will be measured with 'Moxy' muscle oxygenation device during cardiopulmonary exercise test and six-minute walk test. Measurements will be done over quadriceps femoris, locally. Local muscle oxygen saturation and total hemoglobin amount will be assessed during the both tests.
Physical activity level | Second day
  Physical activity level will be evaluated with multi sensor activity device. Patients will be asked to wear the device for five consecutive days on weekdays.
Pulmonary function | Second day
  Dynamic lung volumes and diffusion capacity will be evaluated by using a spirometry according to the American Thoracic Society and European Respiratory Society criteria.
Functional exercise capacity | Second day
  Six-minute walk test will be used to evaluate functional exercise capacity. The test will be done according to American Thoracic Society and European Respiratory Society criteria.
Respiratory muscle strength | Second day
  Respiratory muscle strength will be assessed with mouth pressure device. Maximal inspiratory and expiratory pressure will be measured during the test.
Peripheral muscle strength | Second day
  Quadriceps femoris and shoulder abduction muscle strength will be measured by using hand-held dynamometer.
Inspiratory muscle endurance | Second day
  Inspiratory muscle endurance will be measured incremental threshold loading test, in which patients started an initial load of 30% of maximal inspiratory pressure and test load will be increased with among 10% of maximal inspiratory pressure every 2 minutes.
Functional status | First day
  Functional status of patients after COVID-19 will be evaluated with Post COVID-19 Functional Status Scale (PCFS), which was developed specifically for COVID patients. Limitation and improvement in the functional status of patients after COVID could be assessed with this scale. Functional status were graded from 0 (no functional limitations) to 4 (severe functional limitations) in the scale.
Dyspnea perception | First day
  Dyspnea perception during the daily living activities will be evaluated by using London Chest Daily Living Activity Scale. The highest total score could be obtained from the scale was 75, which indicates significant limitation in daily living activities due to dyspnea perception.
Fatigue | First day
  Fatigue will be assessed with Fatigue Severity Scale (Turkish version). This scale includes 9 items and each item scores from 1 (strong disagreement) to 7 (strong agreement) point. Fatigue Severity Scale total score is calculates by deriving an arithmetic mean. Cut-score of over 4 means significant fatigue and higher score indicates more severe fatigue.
Life Quality | Second day
  Quality of life will be assessed with Saint George Respiratory Questionnaire (SGRQ) (Turkish version). This questionnaire scores range from 0 to 100. The total highest score indicates poor quality of life.
Borg Scale | During exercise training
  Borg Scale will be used to assess dyspnea and fatigue perception of patients during the exercise training. This scale was graded between 6 (no exertion at all) and 20 (maximal exertion).
Modified Borg Scale | During the exercise tests
  Modified Borg Scale will be used to assess dyspnea and fatigue perception of patients during cardiopulmonary exercise training and six-minute walk test. This scale was graded between 0 (nothing at all) and 10 (very very hard).

CONTACTS AND LOCATIONS:
Overall Officials: Ece BAYTOK, MsC, Study Chair — Gazi University; Başak Kavalcı KOL, MsC, Principal Investigator — Gazi University; Nilgün Yılmaz DEMİRCİ, Assoc.Prof, Principal Investigator — Gazi University; Meral Boşnak GÜÇLÜ, Prof. Dr, Study Director — Gazi University
Locations (1):
- Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Clinic, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yao XH, Li TY, He ZC, Ping YF, Liu HW, Yu SC, Mou HM, Wang LH, Zhang HR, Fu WJ, Luo T, Liu F, Guo QN, Chen C, Xiao HL, Guo HT, Lin S, Xiang DF, Shi Y, Pan GQ, Li QR, Huang X, Cui Y, Liu XZ, Tang W, Pan PF, Huang XQ, Ding YQ, Bian XW. [A pathological report of three COVID-19 cases by minimal invasive autopsies]. Zhonghua Bing Li Xue Za Zhi. 2020 May 8;49(5):411-417. doi: 10.3760/cma.j.cn112151-20200312-00193. Chinese. PMID 32172546
- [Result] You J, Zhang L, Ni-Jia-Ti MY, Zhang J, Hu F, Chen L, Dong Y, Yang K, Zhang B, Zhang S. Anormal pulmonary function and residual CT abnormalities in rehabilitating COVID-19 patients after discharge. J Infect. 2020 Aug;81(2):e150-e152. doi: 10.1016/j.jinf.2020.06.003. Epub 2020 Jun 5. No abstract available. PMID 32512021
- [Result] Huang Y, Tan C, Wu J, Chen M, Wang Z, Luo L, Zhou X, Liu X, Huang X, Yuan S, Chen C, Gao F, Huang J, Shan H, Liu J. Impact of coronavirus disease 2019 on pulmonary function in early convalescence phase. Respir Res. 2020 Jun 29;21(1):163. doi: 10.1186/s12931-020-01429-6. PMID 32600344
- [Result] Mo X, Jian W, Su Z, Chen M, Peng H, Peng P, Lei C, Chen R, Zhong N, Li S. Abnormal pulmonary function in COVID-19 patients at time of hospital discharge. Eur Respir J. 2020 Jun 18;55(6):2001217. doi: 10.1183/13993003.01217-2020. Print 2020 Jun. PMID 32381497
- [Result] Raman B, Cassar MP, Tunnicliffe EM, Filippini N, Griffanti L, Alfaro-Almagro F, Okell T, Sheerin F, Xie C, Mahmod M, Mozes FE, Lewandowski AJ, Ohuma EO, Holdsworth D, Lamlum H, Woodman MJ, Krasopoulos C, Mills R, McConnell FAK, Wang C, Arthofer C, Lange FJ, Andersson J, Jenkinson M, Antoniades C, Channon KM, Shanmuganathan M, Ferreira VM, Piechnik SK, Klenerman P, Brightling C, Talbot NP, Petousi N, Rahman NM, Ho LP, Saunders K, Geddes JR, Harrison PJ, Pattinson K, Rowland MJ, Angus BJ, Gleeson F, Pavlides M, Koychev I, Miller KL, Mackay C, Jezzard P, Smith SM, Neubauer S. Medium-term effects of SARS-CoV-2 infection on multiple vital organs, exercise capacity, cognition, quality of life and mental health, post-hospital discharge. EClinicalMedicine. 2021 Jan 7;31:100683. doi: 10.1016/j.eclinm.2020.100683. eCollection 2021 Jan. PMID 33490928